CLINICAL TRIAL: NCT03621683
Title: Antioxidants vs.Ovarian Bio-stimulation Therapy to Rescue the Ovarian Reserve
Brief Title: Antioxidants vs. Ovarian Bio-stimulation Therapy to Rescue the Ovarian Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucy Coleman (Industry)
Responsible Party: Sponsor-Investigator, Lucy Coleman, Scientific director, Fertiaguerrevere
Organization: Fertiaguerrevere (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J298384255
Record Dates: First submitted 2018-07-28; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Reserve

STUDY DESIGN:
Intervention Model Description: Prospective comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ovarian bio-stimulation (Experimental): Intervention:
  ovarian bio-stimulation: blood rich plasma platelets
  Interventions: Procedure: blood rich plasma platelets; Dietary Supplement: Antioxidant therapy
- Antioxidant therapy (Active Comparator): Intervention:
  antioxidants: Q10, DHEA, Vitamin E, Vitamin C, omega 3
  Interventions: Procedure: blood rich plasma platelets; Dietary Supplement: Antioxidant therapy

INTERVENTIONS:
Procedure: blood rich plasma platelets — Injection of blood rich platelet into the ovaries.
Dietary Supplement: Antioxidant therapy — Antioxidants:
  Q10, DHEA, Vitamina E, Vitamin C, Omega 3

SUMMARY:
Two group of patients were selected. Group 1 represents 46 patients that received ovarian-biostimulation monthly for three months. Group 2 represents 32 patients that received antioxidant therapy daily for 3 months. Results are noted and analysed.

Both groups represent patients with procedures already ongoing, and with diagnosed poor or depleted ovarian reserve.

The analysis has been made to compare the efficacy of both procedures.

DETAILED DESCRIPTION:
The bioestimulation group received a blood rich platelet therapy monthly for three months, with a technique developed by the laboratory. The second group of antioxidants received a combination of antioxidants monthly for three months. Both groups were compared to assess the results in terms of ovarian response (number of astral follicles, AMH levels, FSH, LH), and egg quality, embryo development, implantation rate, and successful pregnancy with healthy live birth.

ELIGIBILITY:
Inclusion Criteria:

* Age between 38 and 46 years
* FSH> 12 mIU
* Estradiol > 100 pg/ml
* AMH < 0.8 ng/mL

Exclusion Criteria:

* Pelvic inflammatory syndrome
* vaginal pathologies
* known history of hyperandrogenism
* diagnosed platelet disorders as adhesion
* aggregation
* disorder of thromboxane synthesis.

Ages: 38 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
variation of hormones FSH and LH directly involved with ovarian reserve | 18 months
  Both groups are compared after bio-stimulation and antioxidant therapy is performed to access any possible changes with FSH-LH post-treatment.
variation of AMH directly involved with ovarian reserve in both groups | 18 months
  Both groups are compared after bio-stimulation and antioxidant therapy is performed to access any possible changes with AMH values.
variation in recruitment of antral follicles in both groups | 18 months
  Both groups are compared after bio-stimulation and antioxidant therapy is performed to access any possible changes with the number of astral follicles available.

SECONDARY OUTCOMES:
Number of good quality eggs obtained in both groups after IVF | 18 months
  Egg quality is evaluated in both group of women undergoing IVF after bio-stimulation or antioxidant therapy are performed
Number and quality of fertilised eggs obtained in both groups after IVF | 18 months
  the number and quality of fertilised eggs is evaluated in both groups of women undergoing IVF after bio-stimulation or antioxidant therapy is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Navarro, MD, Principal Investigator — Medical staff
Locations (1):
- Fertiaguerrevere Fertility, Caracas, Disfrito Federal, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided
Still deciding if sharing information. It can be shared as long as it does not contain personal identification such as name, and contact details. We might share the rest of information to other scientist studying the same area of low-depleted ovarian reserve and bio-stimulation techniques.

REFERENCES:
- [Result] Bhartiya D, Parte S, Patel H, Sriraman K, Zaveri K, Hinduja I. Novel Action of FSH on Stem Cells in Adult Mammalian Ovary Induces Postnatal Oogenesis and Primordial Follicle Assembly. Stem Cells Int. 2016;2016:5096596. doi: 10.1155/2016/5096596. Epub 2015 Nov 9. PMID 26635884
- [Result] Telfer EE. Germline stem cells in the postnatal mammalian ovary: a phenomenon of prosimian primates and mice? Reprod Biol Endocrinol. 2004 May 18;2:24. doi: 10.1186/1477-7827-2-24. No abstract available. PMID 15149546
- [Result] Johnson J, Canning J, Kaneko T, Pru JK, Tilly JL. Germline stem cells and follicular renewal in the postnatal mammalian ovary. Nature. 2004 Mar 11;428(6979):145-50. doi: 10.1038/nature02316. PMID 15014492
- [Result] Pan Z, Sun M, Liang X, Li J, Zhou F, Zhong Z, Zheng Y. The Controversy, Challenges, and Potential Benefits of Putative Female Germline Stem Cells Research in Mammals. Stem Cells Int. 2016;2016:1728278. doi: 10.1155/2016/1728278. Epub 2015 Dec 15. PMID 26788065
- [Result] Ozakpinar OB, Maurer AM, Ozsavci D. Ovarian stem cells: From basic to clinical applications. World J Stem Cells. 2015 May 26;7(4):757-68. doi: 10.4252/wjsc.v7.i4.757. PMID 26029346
- [Result] Diamanti-Kandarakis E, Dattilo M, Macut D, Duntas L, Gonos ES, Goulis DG, Gantenbein CK, Kapetanou M, Koukkou E, Lambrinoudaki I, Michalaki M, Eftekhari-Nader S, Pasquali R, Peppa M, Tzanela M, Vassilatou E, Vryonidou A; COMBO ENDO TEAM: 2016. MECHANISMS IN ENDOCRINOLOGY: Aging and anti-aging: a Combo-Endocrinology overview. Eur J Endocrinol. 2017 Jun;176(6):R283-R308. doi: 10.1530/EJE-16-1061. Epub 2017 Mar 6. PMID 28264815
- [Result] Gat I, Blanco Mejia S, Balakier H, Librach CL, Claessens A, Ryan EA. The use of coenzyme Q10 and DHEA during IUI and IVF cycles in patients with decreased ovarian reserve. Gynecol Endocrinol. 2016 Jul;32(7):534-7. doi: 10.3109/09513590.2015.1137095. Epub 2016 Feb 1. PMID 26829445
- [Result] Ozcan P, Ficicioglu C, Kizilkale O, Yesiladali M, Tok OE, Ozkan F, Esrefoglu M. Can Coenzyme Q10 supplementation protect the ovarian reserve against oxidative damage? J Assist Reprod Genet. 2016 Sep;33(9):1223-30. doi: 10.1007/s10815-016-0751-z. Epub 2016 Jun 3. PMID 27255570